CLINICAL TRIAL: NCT03002610
Title: Presenting Summary Information From Cochrane Systematic Reviews to Physicians: Protocol for Research of Infographics Presentation vs. Plain Language Summary
Brief Title: Presenting Summary Information From Cochrane Systematic Reviews to Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Split (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Principal Investigator, Ivan Buljan, Research Assistant, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IP-2014-12-7672
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior | interventions — Cathepsin C

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PLS (Active Comparator): The control group will receive PLS: text format with simple explanation of the survey topic main findings and is intended for lay audience.
  Interventions: Other: Pls
- Infographics (Experimental): Infographics format of a Cochrane systematic review summary represents the experimental intervention in the trial, where the results are presented with text and pictures.
  Interventions: Other: Infographics
- Scientific abstract (Active Comparator): Scientific abstract is the text written for the academic population and practitioners. It is also intended for control group.
  Interventions: Other: Scientific abstract

INTERVENTIONS:
Other: Pls — Text format with simple explanation of the survey topic main findings and is intended for lay audience.
  Arms: PLS
Other: Infographics — Cochrane started developing infographics, where short textual information about research is supported by visual representations of the main findings and is also aimed at the lay public The investigators will examine whether this format is better in information uptake than standard PLS.
  Arms: Infographics
Other: Scientific abstract — Scientific abstract the text written for the academic population and practitioners, with scientific abbreviations which enables experts to go into more detail about the topic.
  Arms: Scientific abstract

SUMMARY:
The objective of this study is to evaluate the efficacy of infographics, compared to standard PLS and scientific abstract format, in presenting information, in terms of understanding and remembering research results by physicians.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial (RCT) with three different formats of the same systematic review summary (Infographics, PLS, scientific abstract). The content of these three formats is based on the same systematic review, but the ways of data presentation will differ: visual presentation in plain language, plain language only, and text with scientific abbreviations. The interventions will be delivered online in January 2016, with physicians who are currently working at Clinical Hospital Split. The trial will be preformed online, and it will be voluntary and anonymous. The survey will consist of 5 parts, in the following order: 1) one format of the summary (randomly assigned), 2) health numeracy, 3) demographic data 4) comprehension test of the information given in the summary, and 5) user friendliness of information and overall satisfaction with the given summary assessed by survey.

ELIGIBILITY:
Inclusion Criteria:

* physicians who are working at Clinical Hospital Split

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Buljan, Principal Investigator — Researcher
Locations (1):
- University of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Osborn CY, Wallston KA, Shpigel A, Cavanaugh K, Kripalani S, Rothman RL. Development and validation of the General Health Numeracy Test (GHNT). Patient Educ Couns. 2013 Jun;91(3):350-6. doi: 10.1016/j.pec.2013.01.001. Epub 2013 Feb 21. PMID 23433635
- See also: Description: Web page where new formats for presentation of Cochrane systematic reviews can be found. — http://visuallycochrane.net

RESULTS

PARTICIPANT FLOW:
Groups:
- Plain Language Summary: The control group will receive PLS: text format with simple explanation of the survey topic main findings and is intended for lay audience.
  Pls: Text format with simple explanation of the survey topic main findings and is intended for lay audience.
Period: Overall Study
Arm/Group | Plain Language Summary | Infographics | Scientific Abstract
Started | 24 | 50 | 34
Completed | 18 | 25 | 21
Not Completed | 6 | 25 | 13
Not completed — Withdrawal by Subject | 6 | 25 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plain Language Summary | Infographics | Scientific Abstract | Total
Number analyzed (Participants) | 18 | 25 | 21 | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40.0 [29.0 to 54.5] | 36.0 [30.0 to 48.5] | 38.0 [29.0 to 48.5] | 37.0 [30.0 to 50.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 16 | 33
  Male | 9 | 17 | 5 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Croatia | 18 | 25 | 21 | 64
Specialization obtained [Count of Participants; unit: Participants] | 13 | 18 | 15 | 46
PhD degree [Count of Participants; unit: Participants] | 9 | 13 | 7 | 29
Heard of Cochrane systematic reviews before [Count of Participants; unit: Participants] | 18 | 23 | 20 | 61
Used Cochrane library [Count of Participants; unit: Participants] | 17 | 17 | 15 | 49

OUTCOME MEASURES:

1. Primary Outcome: Understanding of the Content of Summary Format
Description: The questions will focus on understanding the benefits and risks of the intervention and the quality of evidence described in the systematic review. In total, there will be 10 open ended questions, and the total score will be the sum of the correct answers (minimum 0, maximum 10). Higher scores would indicate higher understanding.
Time Frame: One month (30 days)
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Plain Language Summary | Infographics | Scientific Abstract
Number analyzed (Participants) | 18 | 25 | 21
units on a scale | 8.0 [7.0 to 9.0] | 8.0 [6.0 to 8.0] | 8.0 [5.9 to 9.0]

2. Secondary Outcome: Reading Experience
Description: This section of the survey will include 5 questions about the experience of participants about the text they read, measured on a 10-point Likert type scale, where 1 means do not agree at all and 10 means fully agree. The total score is the sum of scores on all five answers (minimum 5, maximum 50). Higher scores would indicate higher, or more positive, reading experience.
Time Frame: One month (30 days)
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Plain Language Summary | Infographics | Scientific Abstract
Number analyzed (Participants) | 18 | 25 | 21
units on a scale | 32.0 [30.0 to 39.9] | 37.0 [26.8 to 41.3] | 24.0 [21.3 to 31.8]

3. Secondary Outcome: User Friendliness
Description: This section of the survey will have 5 questions concerning how easy it was for the participant to find relevant information, measured by a 10-point Likert type scale where the answer 1 means I do not agree at all and 10 means I fully agree. The total score is the sum of scores on all the answers (minimum 5, maximum 50). Higher scores would indicate greater, or more positive user friendliness, meaning that participants consider that format as easier to find relevant information.
Time Frame: One month (30 days)
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Plain Language Summary | Infographics | Scientific Abstract
Number analyzed (Participants) | 18 | 25 | 21
units on a scale | 29.0 [26.8 to 36.2] | 36.0 [30.9 to 40.0] | 25.0 [23.5 to 27.2]

4. Other Pre Specified Outcome: Health Numeracy
Description: This section will use 6-item General health numeracy test (Osborne et al., 2013) in order to determine how much our participants understand the basic health instructions regarding numeracy dimension. For each correct answer, the participants receive one point and the total score is the sum of all correct answers.
Time Frame: One month (30 days)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Plain Language Summary | Infographics | Scientific Abstract
Number analyzed (Participants) | 18 | 25 | 21
units on a scale | 5.0 [5.0 to 6.0] | 5.0 [4.0 to 6.0] | 5.0 [4.0 to 6.0]

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected.
Description: 0
Arm/Group | Plain Language Summary | Infographics | Scientific Abstract
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor had no role in planning of research, its execution or publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT03002610/Prot_SAP_000.pdf